CLINICAL TRIAL: NCT06189079
Title: Embolizzazione Arteriosa Per il Trattamento Delle Metastasi Ossee: Studio Osservazionale Prospettico
Brief Title: Arterial Embolization for the Treatment of Bone Metastases: Prospective Observational Study
Acronym: EMBONEMET
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: CE AVEC: 313/2023/Oss/IOR
Record Dates: First submitted 2023-11-30; First posted 2024-01-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Bone Metastases
Keywords: Arterial embolization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date, arterial embolization constitutes one of the most popular methods in minimally invasive treatment of bone metastases, allowing good results in terms of pain reduction, local control of disease and reduction of peri-operative bleeding, with low invasiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex of age or older who are candidates for embolization therapy
* Life expectancy > 3 months
* Single metastatic or oligometastatic.
* Plurimetastatic if a particular site is causing painful symptoms or at risk for pathologic rupture

Exclusion Criteria:

* Patients with life expectancy <3 months or severe functional status impairment (ASA 4)
* Patients with hypovascular metastasis documented by angiography or MRI perfusion study with MDC.
* Patients with coagulation deficiency or plateletopenic patients.
* Patients with documented active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent arterial embolization in the treatment of bone metastases
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain (VAS score) | 1 year
  Clinical assessment regarding pain by Visual Analogue Scale (VAS) score (0-100 mm), in which 0 represents no pain, and 100 represents maximum pain imaginable.
Improvement in quality of life (EORTC QLQ - BM22) | 1 year
  Clinical assessment regarding quality of life by EORTC QLQ - BM22 questionnaire. The questionnaire consists of several scales, covering different aspects related to palliation. The maximum and minimum scores for each scale of the questionnaire can range from 0 to 100. The interpretation of scores depends on the specific scale in the questionnaire, and a higher value may indicate either greater negative impact (e.g., more symptoms or more suffering) or greater positive impact (e.g., better quality of life or less symptomatology). The overall assessment requires a detailed analysis of individual scores and related scales.
Improvement in quality of life (EORTC QLQ-C15-PAL questionnaire) | 1 year
  Clinical assessment regarding quality of life by EORTC QLQ-C15-PAL questionnaire. The questionnaire consists of several scales, covering different aspects related to palliation. The maximum and minimum scores for each scale of the questionnaire can range from 0 to 100. The interpretation of scores depends on the specific scale in the questionnaire, and a higher value may indicate either greater negative impact (e.g., more symptoms or more suffering) or greater positive impact (e.g., better quality of life or less symptomatology). The overall assessment requires a detailed analysis of individual scores and related scales.

SECONDARY OUTCOMES:
Volume reduction in cm | 1 year
  Reduction of the lesion evaluated with CT scans, measuring the diameter of the lesion in cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy